CLINICAL TRIAL: NCT01394822
Title: Neuromuscular Ultrasound for Focal Neuropathies
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: NINDS-K23NS062892
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2014-12

CONDITIONS: Focal Neuropathies; Carpal Tunnel Syndrome; Cubital Tunnel Syndrome; Median Neuropathy; Ulnar Neuropathy; Peroneal Neuropathy; Radial Neuropathy; Sciatic Neuropathy; Tibial Neuropathy
MeSH Terms: conditions — Carpal Tunnel Syndrome; Cubital Tunnel Syndrome; Median Neuropathy; Ulnar Neuropathies; Peroneal Neuropathies; Radial Neuropathy; Sciatic Neuropathy; Tibial Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultrasound results reported
- Ultrasound results NOT reported

SUMMARY:
The purpose of this study is to determine if a new diagnostic technique, called neuromuscular ultrasound, can improve our ability to diagnose focal nerve disease.

ELIGIBILITY:
Inclusion Criteria:

* Electrodiagnostic finding of focal nerve disease
* Age 18 and older

Exclusion Criteria:

* Skin lesions preventing ultrasound
* Known ultrasound gel allergy
* Unable to complete 6 months of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals presenting to the Diagnostic Neurology Laboratory at Wake Forest Baptist Medical Center for evaluation of focal nerve disease.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Overall Neuropathy Sum Score | 6 months
  Neuropathy specific scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Cartwright, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Mandeville R, Wali A, Park C, Groessl E, Walker FO, Cartwright MS. Cost-effectiveness of neuromuscular ultrasound in focal neuropathies. Neurology. 2019 Jun 4;92(23):e2674-e2678. doi: 10.1212/WNL.0000000000007602. Epub 2019 May 3. PMID 31053668